CLINICAL TRIAL: NCT01638442
Title: An Open-label, Randomized, Two-way Crossover Trial of the Effect of a High-Fat Meal on the Pharmacokinetics of Oral Tosedostat (CHR 2797) in Healthy Male Subjects
Brief Title: Crossover Trial of the Effect of a High-Fat Meal on the PK of Oral CHR 2797 in Healthy Male Subjects
Acronym: 8265134
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: Chroma Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TST101
Record Dates: First submitted 2012-06-18; First posted 2012-07-11 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Healthy
Keywords: Male subjects, healthy
MeSH Terms: interventions — tosedostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Two 60 mg capsules (120 mg dose) of CHR-2797 administered orally with 240 mL room temperature tap water after an approximately 10 hour fast.
  Interventions: Drug: CHR-2797
- Treatment B (Experimental): Two 60 mg capsules (120 mg dose) of CHR-2792 administered orally with 240 mL room temperature tap water within 30 minutes of receiving a high-fat meal.
  Interventions: Drug: CHR-2797

INTERVENTIONS:
Drug: CHR-2797 — Two 60 mg capsules (120 mg dose) of CHR-2797 administered orally with 240 mL room temperature tap water after an approximately 10 hour fast.
  Arms: Treatment A
Drug: CHR-2797 — Two 60 mg capsules (120 mg dose) of CHR-2792 administered orally with 240 mL room temperature tap water within 30 minutes of receiving a high-fat meal.
  --------------------------------------------------------------------------------
  Arms: Treatment B

SUMMARY:
The objectives of this study are to evaluate the safety and tolerability; and to determine the effect of food on the pharmacokinetics (PK) of CHR-2797 in normal healthy male subjects.

DETAILED DESCRIPTION:
This will be a single center, open-label, 2-arm, 2-way, crossover trial to assess the effect of food on CHR-2797 PK following a single 120 mg dose. Approximately 18 normal, healthy male subjects will be enrolled with at least 12 subjects completing the study. Two 60 mg capsules will be administered for a 120 mg dose of CHR-2797 on Days 1 and 8 with a high-fat meal or in the fasted state according to the randomization schedule. Subjects will be confined at the clinical research unit (CRU) from the time of Period 1 Check-in until Clinic Discharge on Day 3, and will return to the CRU on Day 7 for Period 2 Check-in and remain in the CRU until Study Completion (on Day 10 of Period 2). Blood samples for PK analysis will be collected through 48 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects between 18 and 55 years of age, inclusive.
2. Within BMI range of 18.5 to 29.9 kg/m2, inclusive.
3. In good health, determined by no clinically significant ongoing diseases or other conditions that require medication, and/or any other findings from medical history, physical examination, 12-lead ECG, and vital signs.
4. Clinical laboratory evaluations (including chemistry panel fasted [fasted approximately 10 hours], CBC, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator.
5. Negative test for selected drugs of abuse at Screening (does not include alcohol) and at Check-in (does include alcohol; Appendix A).
6. Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus [anti-HCV], and negative HIV antibody screens (Appendix A);
7. Males will either be sterile or agree to use 1 of the following approved methods of contraception: a male condom with spermicide; a sterile sexual partner; use by female sexual partner of an intrauterine device with spermicide; a female condom with spermicide; contraceptive sponge with spermicide; an intravaginal system (e.g., NuvaRing®), a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives from Check-in (Day -1 of Period 1) until 90 days following Clinic Discharge (Day 10).
8. Able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator).
2. Have a disease or condition that requires daily medication.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (except that appendectomy, hernia repair, and/or cholecystectomy will be allowed).
5. History or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant.
6. History of alcoholism or drug addiction within 1 year prior to Check-in (Day -1 of Period 1).
7. Use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Check-in (Day -1 of Period 1).
8. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 30 days prior to Check-in (Day -1 of Period 1).
9. Use of any prescription medications/products within 14 days prior to Check-in (Day 1 of Period 1), unless deemed acceptable by the Investigator;
10. Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in (Day -1 of Period 1), unless deemed acceptable by the Investigator.
11. Use of alcohol-, grapefruit-, or caffeine-containing foods or beverages within 72 hours prior to Check-in (Day -1 of Period 1), unless deemed acceptable by the Investigator.
12. Poor peripheral venous access.
13. Donation of blood from 30 days prior to Screening through Study Completion, inclusive, or of plasma from 2 weeks prior to Screening through Study Completion, inclusive.
14. Receipt of blood products within 2 months prior to Check-in (Day -1 of Period 1).
15. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety Outcome Measurement | 10 days
  Report adverse events, vital signs, electrocardiograms, and clinical laboratory test.
  Averse events, clinical labs, and other safety variables will be analyzed descriptively for all sujects who recieve at least 1 dose of study drug.
Pharmacokinetic Parameter | 10 days
  For each subject the following PK parameters will be calculated, whevever possible, based on the plasma concentrations of CHR-2797 and its metabolite CHR-79888:
  * Maximum observed concentration (Cmax)
  * time to maximum concentration (t-max)
  * area under the concentration-time curve from Hour 0 to the last measureable concentration (AUC0-t)
  * apparent terminal elimination rate constant
  * apparent terminal elimination half-life

SECONDARY OUTCOMES:
Adverse Events | 10 days
  Adverse events will be summarized by presenting the number and percentages of subjects having any adverse event by MED DRA system organ class and preferred term, relationship to study drug and severity/CTCAE grade. All adverse events will be listed.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stoltz, MD, Principal Investigator — Covance; Simran Singh, MS, GWCPM, Study Chair — CTI BioPharma; Bob Wright, PM, Study Director — Covance; Jack Singer, MD, Study Director — CTI BioPharma
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States